CLINICAL TRIAL: NCT07161739
Title: Vaccination Nudges Project: Behavioural Nudges From Pharmacists to Increase Influenza and Travel Vaccination Uptake: A Pragmatic Randomized Control Trial.
Brief Title: Vaccination Nudges From Pharmacists
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); Mint Health + Drugs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REB25-1205
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Stroke; Influenza Human; Influenza Vaccines; Health Behavior Change; Travel-Related Illness
Keywords: Pragmatic Randomized Control Trial; Policy Trial; Waiver of Consent; Behavioral Nudge
MeSH Terms: conditions — Stroke; Influenza, Human; Travel-Related Illness

STUDY DESIGN:
Intervention Model Description: A two-arm individual-level pragmatic randomized policy trial with two letter dimensions, 1) a letter with an influenza and cardiovascular risk reduction message, and 2) a letter with a travel vaccination benefit message, yielding the following groups:
  Letter with an influenza and cardiovascular risk reduction message Letter with a travel vaccination benefit message
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Influenza and Cardiovascular Risk Reduction (Experimental): Participants randomized to the Influenza Risk Reduction arm will receive a letter encouraging ("nudging") influenza vaccination as an influenza and cardiovascular risk reduction method.
  Interventions: Behavioral: Behavioural Nudge (Influenza Risk Reduction)
- Travel Vaccination Benefit (Experimental): Participants randomized to the Travel Vaccination Benefit arm will receive a letter encouraging ("nudging") travel vaccination as a health benefit by reducing the risk of contracting a travel-related illness.
  Interventions: Behavioral: Behavioural Nudge (Travel Vaccination Benefit)

INTERVENTIONS:
Behavioral: Behavioural Nudge (Influenza Risk Reduction) — A behavioural nudge via mailed letter that discusses the benefits of the influenza vaccine in preventing influenza infection and reducing cardiovascular risk.
  Arms: Influenza and Cardiovascular Risk Reduction
Behavioral: Behavioural Nudge (Travel Vaccination Benefit) — A behavioural nudge via mailed letter that discusses the benefits of travel vaccines in preventing travel-related illnesses.
  Arms: Travel Vaccination Benefit

SUMMARY:
The goal of this individual-level pragmatic randomized policy trial is to learn about the impact of behavioural nudges via mailed letters on increasing influenza and travel vaccination uptake in Alberta, Canada. The primary outcome is the proportion of adults receiving influenza and/or travel vaccination. The secondary outcome is the number of stroke events in the 6 months following vaccination. As such, this research aims to answer two key questions:

1. Do behavioural nudges increase influenza and travel vaccination in Alberta?
2. If yes, is there a decrease in the number of stroke events in the 6 months following vaccination?

The two-arm individual level pragmatic randomized trial design includes two letter dimensions, a letter (a "nudge") with an influenza and cardiovascular risk reduction message and a letter with a travel vaccination benefit message, yielding the following groups:

Letter with an influenza and cardiovascular risk reduction message Letter with a travel vaccination benefit message

DETAILED DESCRIPTION:
Study Population Setting This research project will take place in Alberta, Canada and in partnership with Mint Health and Drugs (Mint Pharmacy), an Alberta-based pharmacy corporation. Participants will be recruited through Mint Pharmacy patient records.

Inclusion Criteria 18 years of age and older by September 1, 2025, and visited a Mint Pharmacy site within 1 year of September 1, 2025.

Study Procedures Sampling Size and Strategy Mint Pharmacy will be sending a letter to all active clients (defined as an adult who filled a prescription at their pharmacy in the last year). The investigators estimate this will be 20,000 clients with 10,000 receiving the influenza vaccine nudge and 10,000 receiving the travel vaccine nudge. This population size will allow the investigators to detect an absolute difference of 2% between the two groups with 80% power and α= 0.05.

Recruitment and Screening Mint Pharmacy analysts will pull the study sample from their patient records, including first and last name, date of birth, and sex. The list of participants will be shared with Alberta Strategy for Patient Oriented Research (AbSPOR) analysts for randomization and data linkage. AbSPOR analysts will share the randomized list of participants, including mailing addresses, with the approved mail vendor to print and mail the appropriate nudge letter that the participant has been randomized to receive. The investigators will stratify be geographic zone (North, Edmonton, Central, Calgary, and South) because of the geographic variation in vaccine uptake.

Intervention The Alberta Government provides free influenza vaccines from October through March annually, which corresponds with peak travel vaccine season. Travel vaccines are typically low cost or covered by private insurance. Vaccines are frequently administered by pharmacists in private pharmacies. As a pragmatic trial, there will be no in-person encounters with patients during the trial. The intervention will be delivered through mailed letters with different messages described below, to be delivered in mid-October 2025. The date of the initial letter will be defined as study baseline.

Arm 1 (Letter with an influenza risk reduction message): This letter will be signed by the pharmacist at the Mint Pharmacy site that the participant accesses and will discuss the benefits of the influenza vaccine in preventing influenza infection and cardiovascular disease risk reduction.

Arm 2 (Letter with travel vaccination benefit message): This letter will be signed by the pharmacist at the Mint Pharmacy site that the participant accesses and will discuss the benefits of travel vaccines in preventing travel related disease, such as evidence that vaccination against Hepatitis A, a common travel vaccination, is 90-95% effective in preventing Hepatitis A infection.

Outcomes Primary outcome: receipt of an influenza and/or travel vaccine on or before March 1, 2026.

Secondary outcome: Number of hospitalizations and emergency department visits for influenza and the number of stroke events on or before September 30, 2026 (6 months following influenza vaccination programs)

Blinding Study researchers will be blind to the participants' group allocation. Participants will not be aware that the communications they receive are part of a research study. Because of this deception, the investigators are requesting a waiver of consent and not attaching a patient information form or informed consent form.

Waiver of Consent

A waiver of consent is necessary both logistically and to limit bias. It is not feasible to obtain informed consent with a sample size n=5190. Additionally, because this study aims to investigate health behaviour, obtaining prior consent alerts participants to the existence of other health messages and may affect their response to the health message they do receive, introducing response bias. Our firm commitment to patient engagement and robust patient engagement plan also reduces participant risk. As per the Tri-Council Policy Statement (TCPS) 2.0, Article 3.7A, alterations to the consent process (including waiver of consent) are appropriate when:

1. The research involves no more than minimal risk to the participant
2. The alteration to consent requirements is unlikely to adversely affect the welfare of participants
3. It is impossible or impractical to carry out the research and to address the research questions properly, given the research design, if the prior consent of participants is required

The proposed study meets the above TCPS 2.0 requirements for alterations to the consent process.

Data Collection Mint Pharmacy analysts will pull the study sample from their patient records, including first and last name, date of birth, and sex. The list of participants will be shared with Alberta Strategy for Patient Oriented Research (AbSPOR) analysts for randomization and data linkage. AbSPOR analysts will share the randomized list of participants, including mailing addresses, with the approved mail vendor to print and mail the appropriate nudge letter that the participant has been randomized to receive. AbSPOR analysts will gather vaccination data from the Alberta Health Immunization and Adverse Reactions Following Immunization (IMM/ARI) database by linking participant health numbers to determine how many participants received a vaccination. The IMM/ARI database is the most comprehensive vaccination database as it is where all vaccinations are required to be reported in Alberta with nearly 100% coverage. AbSPOR analysts will gather hospitalization, emergency department visit, and the number of stroke events from the Alberta Health Discharge Abstract Database (DAD) using participant health numbers. Influenza and stroke events will be identified using ICD-10 codes. This data collection will be continuous from April 1st, 2026, through September 30th, 2026, six-months following the influenza vaccination program. Data linkage and cross-reference will be conducted by AbSPOR, who will share de-identified data with the research team in either de-identified or aggregate form for analysis.

Data Analysis Data analysis will be conducted by members of the research team using the de-identified data provided by AbSPOR. Statistical comparisons will be performed according to the intention-to-treat principle. The investigators will report the proportion of adults who received influenza vaccination and travel vaccination (any vaccines, specific vaccine types, and full series of vaccines) in each group along with 95% confidence intervals. The investigators will model the risk difference for each type of nudge compared to the comparison group) in separate models, including adjustment for multiple comparisons. As a secondary analysis, the investigators will assess time to vaccination in the influenza letter group compared to the travel vaccine letter group. To assess impact of vaccine uptake on influenza and stroke events, the investigators will compare the number of events in one intervention group with the number of stroke events in the comparison group. The primary analysis will be conducted on the as-randomized populations (intention-to-treat analysis).

ELIGIBILITY:
Inclusion Criteria:

* Visited a Mint Pharmacy site within 1 year of enrollment date
* 18 years of age and older by enrolment date

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Influenza and/or Travel Vaccination | From enrollment and randomization to the end of the intervention window at 6 months post-enrollment/randomization.
  The proportion of participants who received an influenza and/or travel vaccination.

SECONDARY OUTCOMES:
Stroke Events | From date of vaccination to the end of follow-up at 6 months post-vaccination.
  Number of stroke events among participants in the 6 months following vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Amity Quinn, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Public Health Agency of Canada, Statement on Seasonal Influenza Vaccine for 2014-2015. 2014, National Advisory Committee on Immunization: Ottawa.
- [Background] McAlister FA, Straus SE, Sackett DL, Altman DG. Analysis and reporting of factorial trials: a systematic review. JAMA. 2003 May 21;289(19):2545-53. doi: 10.1001/jama.289.19.2545. PMID 12759326
- [Background] Renosa MDC, Landicho J, Wachinger J, Dalglish SL, Barnighausen K, Barnighausen T, McMahon SA. Nudging toward vaccination: a systematic review. BMJ Glob Health. 2021 Sep;6(9):e006237. doi: 10.1136/bmjgh-2021-006237. PMID 34593513
- [Background] Patel MS, Milkman KL, Gandhi L, Graci HN, Gromet D, Ho H, Kay JS, Lee TW, Rothschild J, Akinola M, Beshears J, Bogard JE, Buttenheim A, Chabris C, Chapman GB, Choi JJ, Dai H, Fox CR, Goren A, Hilchey MD, Hmurovic J, John LK, Karlan D, Kim M, Laibson D, Lamberton C, Madrian BC, Meyer MN, Modanu M, Nam J, Rogers T, Rondina R, Saccardo S, Shermohammed M, Soman D, Sparks J, Warren C, Weber M, Berman R, Evans CN, Lee SH, Snider CK, Tsukayama E, Van den Bulte C, Volpp KG, Duckworth AL. A Randomized Trial of Behavioral Nudges Delivered Through Text Messages to Increase Influenza Vaccination Among Patients With an Upcoming Primary Care Visit. Am J Health Promot. 2023 Mar;37(3):324-332. doi: 10.1177/08901171221131021. Epub 2022 Oct 4. PMID 36195982
- [Background] Modin D, Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Claggett BL, Dueger EL, Samson SI, Loiacono MM, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Jean-Marie Martel C, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Effect of Electronic Nudges on Influenza Vaccination Rate in Older Adults With Cardiovascular Disease: Prespecified Analysis of the NUDGE-FLU Trial. Circulation. 2023 May 2;147(18):1345-1354. doi: 10.1161/CIRCULATIONAHA.123.064270. Epub 2023 Mar 5. PMID 36871213
- [Background] Johansen ND, Vaduganathan M, Bhatt AS, Lee SG, Modin D, Claggett BL, Dueger EL, Samson SI, Loiacono MM, Kober L, Solomon SD, Sivapalan P, Jensen JUS, Martel CJ, Valentiner-Branth P, Krause TG, Biering-Sorensen T. Electronic nudges to increase influenza vaccination uptake in Denmark: a nationwide, pragmatic, registry-based, randomised implementation trial. Lancet. 2023 Apr 1;401(10382):1103-1114. doi: 10.1016/S0140-6736(23)00349-5. Epub 2023 Mar 5. PMID 36889332
- [Background] Saaksvuori L, Betsch C, Nohynek H, Salo H, Sivela J, Bohm R. Information nudges for influenza vaccination: Evidence from a large-scale cluster-randomized controlled trial in Finland. PLoS Med. 2022 Feb 9;19(2):e1003919. doi: 10.1371/journal.pmed.1003919. eCollection 2022 Feb. PMID 35139082
- [Background] Holodinsky JK, Zerna C, Malo S, Svenson LW, Hill MD. Association between influenza vaccination and risk of stroke in Alberta, Canada: a population-based study. Lancet Public Health. 2022 Nov;7(11):e914-e922. doi: 10.1016/S2468-2667(22)00222-5. PMID 36334607
- [Background] Yu AYX, Krahn M, Austin PC, Rashid M, Fang J, Porter J, Vyas MV, Bronskill SE, Smith EE, Swartz RH, Kapral MK. Sex differences in direct healthcare costs following stroke: a population-based cohort study. BMC Health Serv Res. 2021 Jun 29;21(1):619. doi: 10.1186/s12913-021-06669-w. PMID 34187462
- [Background] Holodinsky JK, Lindsay P, Yu AYX, Ganesh A, Joundi RA, Hill MD. Estimating the Number of Hospital or Emergency Department Presentations for Stroke in Canada. Can J Neurol Sci. 2023 Nov;50(6):820-825. doi: 10.1017/cjn.2022.338. Epub 2022 Dec 20. PMID 36536997
- [Background] Molinari NA, Ortega-Sanchez IR, Messonnier ML, Thompson WW, Wortley PM, Weintraub E, Bridges CB. The annual impact of seasonal influenza in the US: measuring disease burden and costs. Vaccine. 2007 Jun 28;25(27):5086-96. doi: 10.1016/j.vaccine.2007.03.046. Epub 2007 Apr 20. PMID 17544181
- [Background] Schanzer DL, Sevenhuysen C, Winchester B, Mersereau T. Estimating influenza deaths in Canada, 1992-2009. PLoS One. 2013 Nov 27;8(11):e80481. doi: 10.1371/journal.pone.0080481. eCollection 2013. PMID 24312225
- See also: Alberta Government. Alberta Influenza Statistics. 2023. [cited 2023 May 25]; — https://www.alberta.ca/stats/dashboard/respiratory-virus-dashboard.htm